CLINICAL TRIAL: NCT03629795
Title: Serum Sample Collection to Determine Analytical Performance Characteristics of the ADVIA CENTAUR® PREGNANCY ASSOCIATED PLASMA PROTEIN A and ADVIA Centaur® Free Beta Human Chorionic Gonadotropin ASSAYS
Brief Title: Serum Sample Collection to Determine Analytical Performance Characteristics of the ADVIA Centaur PAPPA and BhCG Assays
Status: Completed | Type: Observational
Sponsor: Axis Shield Diagnostics Ltd (Industry)
Collaborators: The Clinical Trial Company (Industry)
Responsible Party: Sponsor
Other Study IDs: TO06
Record Dates: First submitted 2018-07-26; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Trisomy 21 in Fetus; Trisomy 18 in Fetus; Trisomy 13 in Fetus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Blood samples collected will be shipped to the sponsor's laboratory to establish analytical performance characteristics of the ADVIA Centaur® Pregnancy Associated Plasma Protein A (PAPP-A) and ADVIA Centaur® Free Beta Human Chorionic Gonadotropin (Free βhCG) assays.

DETAILED DESCRIPTION:
Blood samples are to be collected from pregnant women attending their scheduled 1st Trimester scan; the samples are to be collected immediately after the subject's routine blood sample at the clinic visit. No extra venepuncture will be required.

Blood samples collected will be shipped to the sponsor's laboratory to establish analytical performance characteristics of the ADVIA Centaur® Pregnancy Associated Plasma Protein A (PAPP-A) and ADVIA Centaur® Free Beta Human Chorionic Gonadotropin (Free βhCG) assays.

ELIGIBILITY:
Inclusion Criteria:

* A subject is considered eligible for participation in the trial if all of the following inclusion criteria are satisfied prior to enrolment:

  1. Subject is ≥ 18 years of age
  2. Subject is informed and has been given ample time and opportunity to think about her participation and has given her written informed consent.
  3. Women with a structurally normal viable pregnancy with a fetal crown rump length of 45-84 mm

Exclusion Criteria:

* A subject is not eligible for participation in the trial if any of the following exclusion criteria are met prior to enrolment:

  1. Subject is unable to give consent
  2. Subject has already participated in the study

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: First trimester pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Sample handling | 3 months
  Percentage change in PAPPA and BhCG levels from baseline sample type to sample type under test.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Robson, Principal Investigator — Professor of Fetal Medicine
Locations (1):
- Newcastle University, Newcastle upon Tyne, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No